CLINICAL TRIAL: NCT01769872
Title: Safety and Effect of Adipose Tissue Derived Mesenchymal Stem Cell Implantation in Patients With Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: R-Bio (Industry)
Collaborators: Korea University Anam Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSC-MSCs-SPI
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

ARMS (1):
- Autologous Adipose Tissue derived MSCs (Experimental)
  Interventions: Procedure: Autologous Adipose Tissue derived MSCs Transplantation

INTERVENTIONS:
Procedure: Autologous Adipose Tissue derived MSCs Transplantation — Intravenous injection of Autologous Adipose Derived Mesenchymal Stem Cells. Dose : 2x10e8 cells / 20mL Intrathecal injection of Autologous Adipose Derived Mesenchymal Stem Cells. Dose : 5x10e7 cells / 2mL Into a spinal cord injection of Autologous Adipose Derived Mesenchymal Stem Cells. Dose : 2x10e7 cells / 1mL

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of autologous transplantation of Adipose Tissue derived Mesenchymal stem cells (MSCs) in patient with spinal cord injury

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and sign the consent form for this study
* Age : 19-70
* Clinical diagnosis of spinal cord injury(American Spinal Injury Association[ASIA] Impairment Scale[AIS] grade A or B or C)
* Duration of injury : > 3 month

Exclusion Criteria:

* Subjects who must put on a respirator
* Subjects who had malignant tumor within 5 years
* Subjects with a infectious disease include HIV and hepatitis
* Subjects who injured brain or spinal cord before spinal cord injury
* Subjects with anemia or thrombocytopenia
* Subjects with angina pectoris, myocardial infarction, cardiomyopathy, occlusive disease, chronic renal failure, glomerular disease and chronic obstructive pulmonary disease
* Subjects with congenital or acquired immunodeficiency disorders
* Patients with clouded consciousness or speech disorder
* treat with cytotoxic medications(immunosuppressive drug, corticosteroid and cytotoxic drug) during clinical trials
* participating another clinical trials within 3 months
* other serious disease or disorder that could seriously affect ability to participate in the study

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
ASIA (American Spinal Injury Association) scale | 32 weeks
  To evaluate the change of treated spinal cord before cell implantation and at 3 and 6 months post injection of MSCs.

SECONDARY OUTCOMES:
Magnetic Resonance Imaging | 32 weeks
  To evaluate the change of treated spinal cord injury using Magnetic Resonance Imaging (MRI) at 3 and 6 months post injection of MSCs.
MEP/SSEP | 32 weeks
  To evaluate the change of treated spinal cord before cell implantation and at 3 and 6 months post injection of MSCs.
ADL (activities of daily living) | 32 weeks
  To evaluate the change of treated spinal cord before cell implantation and at 3 and 6 months post injection of MSCs.
SF-36 | 32 weeks
  To evaluate the change of treated spinal cord before cell implantation and at 3 and 6 months post injection of MSCs.
ODI (Oswestry Disability Questionnaire) | 32 weeks
  To evaluate the change of treated spinal cord before cell implantation and at 3 and 6 months post injection of MSCs.
Frequency of Adverse Events | 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Hyoung Cho, M.D. & Ph.D., Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea